CLINICAL TRIAL: NCT05475080
Title: Carotid Web and Stroke Registry. Clinical and Genetic Study. "Registro de Pacientes Con Carotid Web e Ictus. Estudio clínico y genético"
Brief Title: Carotid Web and Stroke Registry.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Other Study IDs: IIBSP-CWI-2022-33
Record Dates: First submitted 2022-07-22; First posted 2022-07-26 (Actual); Last update posted 2022-08-01 (Actual); Status verified 2022-07

CONDITIONS: Stroke; Carotid Web
MeSH Terms: conditions — Stroke | interventions — Platelet Aggregation Inhibitors; Anticoagulants; Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Antiplatelet
  Interventions: Drug: Antiplatelet Drug
- Anticoagulant
  Interventions: Drug: Anticoagulant
- Endovascular
  Interventions: Procedure: Endovascular
- Surgical (endarterectomy)
  Interventions: Procedure: Surgery

INTERVENTIONS:
Drug: Antiplatelet Drug — Any antiplatelet drug or combination
  Groups: Antiplatelet
Drug: Anticoagulant — Any anticoagulante
  Groups: Anticoagulant
Procedure: Endovascular — Angioplasty +- stent
  Groups: Endovascular
Procedure: Surgery — Endarterectomy
  Groups: Surgical (endarterectomy)

SUMMARY:
Introduction:

Carotid Web (CW) is a common cause of stroke in young patients with a high recurrence rate. The factors associated with recurrences and the appropriate treatment to prevent them are currently unknown.

Main objective:

To compare recurrences of ischemic stroke (cerebral infarction or transient ischemic attack) in patients with CW according to the preventive treatment.

Secondary objectives:

* To describe the frequency of recurrences in patients with stroke and CW.
* To compare the risk of complications, especially hemorrhagic complications, in patients with stroke and CW according to the type of preventive treatment given.
* To describe the clinical and radiological characteristics of CW and identify which are associated with recurrences.
* To detect genetic polymorphisms associated with the presence of CW in stroke patients.

Study design:

Multicenter, prospective registry of consecutive cases with ischemic stroke in which a Carotid Web is detected between 2022 and 2024.

All patients with ischemic stroke or transient ischemic attack and age > or = 18 years, in whom a Carotid Web is diagnosed, will be included. Demographic and clinical variables, genetic study (not mandatory), diagnostic methods of CW, reperfusion treatment and secondary prevention will be collected. During a minimum follow-up of six months, vascular events (stroke, transient ischemic accidents, cerebral hemorrhages) and treatments (antiplatelet therapy, anticoagulation, endarterectomy, endovascular therapy) will be collected.

Once the registry has been completed, the frequency of recurrences and the factors associated with them will be analyzed.

Study population:

Patients with ischemic stroke or transient ischemic attack in whom a Carotid Web is detected. It is estimated to obtain data from approximately 100 patients.

Variables:

Demographic, clinical (past medical history, stroke characteristics), radiological (diagnostic method of CW, morphological characteristics of CW), therapeutic (preventive treatment initiated) and prognostic variables will be collected. Recurrences in the form of stroke or transient ischemic attack (main variable) will be collected during a minimum follow-up of six months. Cerebral hemorrhages, mortality and therapeutic changes during follow-up will also be collected.

Ethical considerations:

This is an observational registry, with no changes in the management or treatment of the patients included, and with an anonymized data registry. Written informed consent will be requested from the patient or his/her representative for participation in the registry and for obtaining a blood sample for the genetic study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ischemic stroke or TIA and
* Age > or = 18 years.
* Carotid Web diagnosed by angioCT, angioMRI or arteriography.
* Consent to participate from patient or representative

Exclusion Criteria:

* No informed consent obtained

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with ischemic stroke or TIA and an age > or = 18 years, in whom a CW is diagnosed during the etiological study, will be included.
  A CW will be defined by the presence of a focal and homogeneous intraluminal protrusion (shelf-like), without calcific component, located in the posterior or postero-lateral wall of the proximal internal carotid artery or carotid bulb. The diagnosis should be made by angioCT, angioMRI or arteriography.
  Both patients with a CW ipsilateral to the ischemic event and those with a CW unrelated to the ischemic event will be included.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-07-15 (Actual); Primary Completion 2024-07-15 (Estimated); Study Completion 2025-07-15 (Estimated)

PRIMARY OUTCOMES:
Ischemic Recurrences | At least 6 months of follow-up
  Stroke or TIA

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de la Santa Creu i Sant Pau, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes